CLINICAL TRIAL: NCT07145229
Title: A Randomized, Double-blind, Multicenter, Colchicine and Placebo-controlled Study to Evaluate the Efficacy and Safety of ABP-745 in Subjects With an Acute Gout Flare
Brief Title: Safety and Efficacy of ABP-745 in Participants With an Acute Gout Flare
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-745-201
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Gouty Arthritis; Gout Flare; Gout Flares; Acute Gout Flare
Keywords: Gout; Gout Flare; Colchicine; Acute gout flare; ABP-745
MeSH Terms: conditions — Gout | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABP-745 Dose A (Experimental)
  Interventions: Drug: ABP-745 Dose A
- ABP-745 Dose B (Experimental)
  Interventions: Drug: ABP-745 Dose B
- Colchicine (Active Comparator)
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABP-745 Dose A — ABP-745 Dose A + Colchicine placebo - tablets (PO)
  Arms: ABP-745 Dose A
Drug: ABP-745 Dose B — ABP-745 Dose B + Colchicine placebo - tablets (PO)
  Arms: ABP-745 Dose B
Drug: Colchicine — ABP-745 placebo + Colchicine - tablets (PO)
  Arms: Colchicine
Drug: Placebo — ABP-745 placebo + Colchicine placebo - tablets (PO)
  Arms: Placebo

SUMMARY:
A randomized, double-blind, international multicenter, colchicine and placebo-controlled study to evaluate the efficacy and safety of ABP-745 in subjects with acute gout. Efficacy of ABP-745 in reducing pain and swelling compared with standard colchicine treatment and placebo will be evaluated in participants with acute gout. The primary efficacy measurement will be pain score after treatment.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects are eligible for the study if they meet all of the following Inclusion Criteria:

* Age 18-70 years old (inclusive), male or female.
* Body mass index (BMI)18-40 kg/m2 (inclusive).
* Medical history and current findings consistent with diagnosis of gouty arthritis.
* Subjects must have experienced 2 or more gout flares within 12 months prior to screening.
* Onset of an acute gout flare, within 6 months
* Patients receiving ULT agents (such as allopurinol, febuxostat, probenecid, etc.) must be on stable doses of these drugs prior to first dose of study drug (and remain on the same dose throughout the Treatment Period).
* Subjects agree to maintain a stable lifestyle (such as diet and exercise) during the study period.

Key Exclusion Criteria:

Subjects are excluded from the study if one or more of the following criteria are met:

* Administration of oral prednisone ≥ 10 mg or equivalent doses of other glucocorticoids, or use of narcotics, within 24 hours prior to first dose of study drug, or intramuscular, intravenous, or intra-articular injection of any glucocorticoid within 14 days prior to first dose of study drug.
* Use of Nonsteroidal Anti-inflammatory Drugs (NSAIDs) prior to first dose dose of study drug, at the investigator's discretion.
* Administration of colchicine or ABP-745 within 14 days prior to first dose of study drug.
* Subjects took any investigational drug in any clinical study within 1 month prior to first dose of study drug and throughout the study period.
* Administration of pegloticase, or methotrexate, or any biologic IL-1 blocker, TNF inhibitor, or other biological agent within 30 days prior to first dose of study drug or within 5 half-lives of the study drug prior to the first dose of study drug, whichever is longer.
* Administration of muscle relaxants, central stimulants, barbiturates, etc. within 30 days prior to first dose of study drug or within 5 half-lives of the drug prior to the first dose of study drug, whichever is longer.
* Secondary gout (e.g., gout induced by chemotherapy, transplant-related gout).
* Subjects with a current diagnosis or history of rheumatoid arthritis, psoriatic arthritis, evidence or suspicion of infectious/septic arthritis, calcium pyrophosphate (CPP) crystal arthritis, acute polyarticular gout (4 or more joints), multiple sclerosis or any other demyelinating disease, or; major chronic inflammatory disease or connective tissue disease other than RA or psoriatic arthritis (PsA), including but not limited to fibromyalgia or systemic lupus erythematosus (with the exception of secondary Sjögrens syndrome, etc.); with arthritis due to any cause other than gout that may confound any study assessments per Investigator discretion or Prosthetic joint infection within 5 years of screening, or native joint infection within 1 year of screening
* Current anticoagulation therapy, thrombocytopenia, or diseases with a risk of thrombocytopenia, such as aplastic anemia, hypersplenism, or known hemorrhagic diseases like idiopathic thrombocytopenic purpura or hemophilia.
* History of malignancy within 5 years prior to screening, excluding localized cancers such as basal cell carcinoma.
* Presence of significant diseases, including but not limited to: uncontrolled hypertension (systolic blood pressure ≥160 or diastolic blood pressure ≥100 mmHg), congestive heart failure (New York Heart Association [NYHA] class III or above), uncontrolled type 1 or 2 diabetes mellitus (hemoglobin A1c [HbA1c] >8.5%). Inclusion will be determined by the Investigator based on the subject's specific condition.
* Women of childbearing potential as defined by Appendix 2.
* Experienced only no or mild gout-related pain prior to first dose of study drug.
* Use of gout flare prophylaxis (e.g., colchicine, NSAIDs, prednisone/methylprednisolone) at the time of randomization based on conversation with subject and self-reported.
* Corona Virus Disease (COVID) vaccination in the 4 weeks prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) pain score of the target joint | 24 hours post the first dose of study drug
  Change from baseline in 0-100 mm VAS pain score of the target joint

SECONDARY OUTCOMES:
Change and percentage change from baseline in VAS pain score of the target joint | 2-8 days post the first dose of study drug
Incidence of treatment-emergent adverse events (Safety and Tolerability) | up to 14 days post the first dose of study drug
  TEAEs and SAEs, and clinically significant changes in physical examination, vital signs, safety laboratory tests, and 12-lead ECG.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (14):
  - Onyx Clinical Research, Peoria, Arizona
  - Exinia Research, La Mesa, California
  - Evergreen Clinical Trial, Norcross, Georgia
  - Bioluminux Clinical Research, Naperville, Illinois
  - Exinia Research, Des Moines, Iowa
  - Northshore Research Associates, Alexandria, Louisiana
  - DelRicht Research, Baton Rouge, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Interphase Clinical Trials, Lutherville, Maryland
  - DelRicht Research Gulfport, Gulfport, Mississippi
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - West Clinical Research, Morehead City, North Carolina
  - DelRicht Research, Tulsa, Oklahoma
  - Premier Family Physicians, Austin, Texas
- Australia (6):
  - Emeritus Sydney, Botany, New South Wales
  - Canopy Clinical Research Northern Beaches, Brookvale, New South Wales
  - Novatrials, Kotara, New South Wales
  - Genesis Research Services, Newcastle, New South Wales
  - Emeritus Melbourne, Camberwell, Victoria
  - Canopy Clinical Research Altona North, North Altona, Victoria
- China (18):
  - Peking University Third hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The second affiliated hospital of guangxi medical university, Nanning, Guangxi
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Wuhan UHospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Xiangya Hospital Zhuzhou Central South University, Zhuzhou, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Linfen Central hospital, Linfen, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Xi'an Daxing Hospital, Xi’an, Shanxi
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided